CLINICAL TRIAL: NCT02413749
Title: DC-STAMP and TRAF3: Regulators of Osteoclastogenesis and Biomarkers in Psoriatic Arthritis
Brief Title: DC-STAMP & TRAF3: Regulators of Osteoclastogenesis and Biomarkers in PsA
Acronym: Incubator
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Christopher Ritchlin, M.D., M.P.H.; Professor of Medicine, Chief of Allergy, Immunology & Rheumatology Division, University of Rochester
Other Study IDs: RSRB 53086
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples that remain after study assays are completed may be stored for future non-genetic research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stable PsA response to treatment: Individuals with psoriatic arthritis who are being treated standard of care with a stable DMARD or a biologic
- PsA inadequate response to DMARD: Individuals with psoriatic arthritis who have had an inadequate response to a DMARD and are being treated standard of care with a biologic.

SUMMARY:
Biologics such as anti-Tumor Necrosis Factor or TNF inhibitor (TNFi) for treatment of Psoriatic Arthritis (PsA) has greatly reduced bone damage. This collaborative study will provide insights into key mechanisms that underlie inflammatory arthritis and bone damage in psoriatic joints and will catalyze biomarker discovery, identifying early biologic responders to facilitate optimization of therapy.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA), an inflammatory joint disease associated with psoriasis (Ps), affects approximately 650,000 adults in the United States and is associated with increased morbidity and mortality. Bone damage develops in half these patients within the first two years of disease, often leaving them with impaired function and diminished quality of life. The emergence of anti-Tumor Necrosis Factor therapies (TNFi) has dramatically improved clinical response and slowed bone and cartilage degradation in PsA patients, however, only 50-60% of patients respond to these agents. To improve these outcomes, investigators must address two major gaps: a limited understanding of key events that underlie pathologic bone destruction and the absence of biomarkers to predict TNFi response and identify early TNFi responders to facilitate optimization of therapy.

Bone damage is mediated by osteoclasts which arise from monocyte precursors in the blood. Osteoclast Precursors (OCPs) are dramatically increased in PsA, compared to controls, particularly in patients with bone damage on X-ray. The number of these circulation precursor cells dropped rapidly following treatment with TNFi. OCPs may serve as response biomarkers, but cost, time and high variability limit these assays. Osteoclast precursors express Dendritic Cell-Specific Transmembrane Protein (DC-STAMP), which is a seven-pass transmembrane protein required for fusion of monocytes to form osteoclasts and giant cells. Monocyte DC-STAMP levels dropped rapidly following treatment with TNFi. TNF receptor-associated factor 3 (TRAF3), an inhibitor of OC formation that correlates with extracellular TNF concentrations, is elevated in OCPs from PsA patients. These markers may predict TNFi treatment response.

The goal of this study is to examine Psoriatic Arthritis patients prior to and after standard of care biologic treatment such as TNFi, while also examining DC-STAMP and TRAF3 expression in a cross-sectional analysis of patients on stable oral disease modifying agents (DMARDS) and in patients in low disease activity state on TNFi therapy.

* Research Assays:

The correlation between TRAF3 and DC-STAMP expression at the RNA and protein level may be examined for two baseline PsA patients by real-time PCR, flow cytometry and western after Chloroquine (CQ) blockade, which prevents TRAF3 degradation. Cells isolated from human PBMC may be sterile sorted prior to use in some in vitro assays. Sorted cells may be treated with CQ or MG132, a proteasome inhibitor, in OC-promoting media in time course and dose-response experiments and OCs counted to determine if DC-STAMP is degraded by the lysosome or proteasome.

Peripheral Blood Mononucleated Cells (PBMCs) will be isolated from blood by centrifugation. These cells may be used for flow cytometry to analyze TRAF3 and DC-STAMP expression on monocytes along with OC quantification at baseline and/or approximately 4 months of treatment. DC-STAMP surface expression on PBMC from PsA patients correlated with the number of OCP in culture and the level of DC-STAMP on CD14+ monocytes declined significantly in PsA patients following TNFi. The decline in DC-sTAMP+CD14+ cells may serve as a measure of early response to TNFi.

ELIGIBILITY:
Inclusion Criteria:

* All Subjects

  1. Ability to provide written informed consent.
  2. Subjects can be of either gender but must be at least 18 years old.
  3. Subjects with PsA should fulfill CASPAR criteria
* Longitudinal

  1. Patients with active PsA starting standard of care biologic treatment.
* Additional Blood Draw

  1. Positive DC-STAMP signal at baseline
* Cross-Sectional 1. Patients on stable DMARDS or biologics for more than 16 weeks.

Exclusion Criteria:

1. Unable to donate blood because of poor venous access or intolerance of phlebotomy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects that are 18 years old and older. Due to the demographic distribution of the disease we expect all or nearly all subjects to be caucasian, however no subjects will be excluded based on race or ethnic origin.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Examination of molecular mechanisms underlying DC-STAMP and TRAF3 mediated osteoclastogenesis | week 0 to week 16
  Investigators will analyze TRAF3 and DC-STAMP expression in monocytes from PsA patients cross-sectionally by flow cytometry. Disease Activity Score 66/68 (DAS66/68), TRAF3 levels and the change in DC-STAMP+CD14+ will be observed to see if they correlate with standard of care treatment.

SECONDARY OUTCOMES:
Assessment of DC-STAMP and TRAF3 as biologic predictor and treatment response markers in PsA | week 0 to week 16
  Investigators will analyze TRAF3 and DC-STAMP expression in monocytes from PsA patients longitudinally by flow cytometry. Disease Activity Score 66/68 (DAS66/68), TRAF3 levels and the change in DC-STAMP+CD14+ will be observed to see if they correlate with standard of care treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD/MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Information of any type may be shared with researchers at other institutions. Subjects will be made aware of this in the informed consent form.
Time Frame: Once a subject signs the consent form to allow for sharing, If any samples remain after all tests are completed, the samples will be stored for future research indefinitely or until the subject cancels consent to share.
Access Criteria: Only investigators that the study team collaborates with will have access to samples. Data will not include any information that is identifying.